CLINICAL TRIAL: NCT03872869
Title: Tai Chi and Hip School for Patients With Hip-OA: a Randomized Controlled Trial With a 6 - and 12 Months Follow-up
Brief Title: Tai Chi and Hip School for Patients With Hip-OA.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anne Sunden, RPT, PhD, Lecturer, Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 73/2005
Record Dates: First submitted 2019-02-25; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; patient education; Tai Chi; physical function
MeSH Terms: conditions — Osteoarthritis | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: After an advertisement in a local paper, over 300 volunteers applied to participate in the study. All 300 received information about the study by mail or telephone. One hundred volunteers fulfilled the inclusion criteria: X-ray-verified hip OA, 40-75 years of age, no walking aid and no joint replacements in the hips or knees. Each individual had to specify at which hospital and when they had been X-rayed and/or received their diagnosis. A total of 89 subjects attended the baseline appointment and were randomized to one of the three groups. The randomization procedure, in blocks of 15, was generated by a computer-based system
Who Masked: Investigator
Masking Description: The investigators did not know which group the patients had been assigned to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hip School (Active Comparator): The participants in the Hip School were required to attend three 1.5 hour classes which were conducted by specially trained physiotherapists in premise at Lund University.
  Interventions: Other: Hip school or Tai CHi for arthritis
- Tai Chi for arthritis (TCA) (Active Comparator): The treatment intervention with TCA was scheduled in a group setting. Class size for Tai Chi groups was 8- 10 individuals. The group was led by a physiotherapist, specially trained in the concept, in premise at Lund University. The participants in the Tai Chi group were required to attend classes for 12-16 one- hour sessions, twice a week for the first four weeks and then once a week.
  Interventions: Other: Hip school or Tai CHi for arthritis
- Control group (No Intervention)

INTERVENTIONS:
Other: Hip school or Tai CHi for arthritis — Eighty-nine individuals were randomized to one of the three intervention groups 30 individuals to Tai Chi,30 individuals to Hip School and 29 individuals to the control group
  Arms: Hip School; Tai Chi for arthritis (TCA)

SUMMARY:
A randomized, controlled study was conducted in southern Sweden with two intervention programs for individuals with X-ray-verified hip osteoarthritis (OA). The patients were randomized to 1 of 3 groups; namely Hip School, Tai Chi for Arthritis (TCA), or a group receiving no intervention. The results showed significant improvement in physical function and self-efficacy within the interventions groups Tai Chi and Hip School. The Tai Chi group showed improvement in body awareness and quality of movements, and in self-efficacy between baseline and 6- month follow-up. The Hip School group showed significant improvement in body awareness and quality of movements between baseline and 6-month follow-up.

DETAILED DESCRIPTION:
A randomized, controlled study was conducted in southern Sweden with two intervention programs for individuals with X-ray-verified hip OA. The patients were randomized to 1 of 3 groups; namely Hip School, TCA, or a group receiving no intervention. A total of 89 subjects attended the baseline appointment and were randomized to one of the three groups. Physical function was assessed using, the Hip Osteoarthritis Outcomes Score (HOOS, Swedish version L.K 1.1), an observational assessment of movements the Body Awareness Scale Movement Quality (BAS MQ) and the Six Minute Walk Test (6MWT). For assessment of HRQL the Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) was used. The Arthritis Self-Efficacy Scale (ASES) records the patient's self-reported judgment of what he/she can do regardless of the degree of functional limitations or skill. Six months after the final intervention all subjects were examined and assessed following the same procedure as at baseline. The 12 months follow-up contained the three questionnaires, HOOS, ASES and SF- 36 were sent out by mail. The results showed significant improvement in physical function and self-efficacy within the interventions groups Tai Chi and Hip School. The Tai Chi showed improvement in BAS MQ, focusing on body awareness and quality of movements, and in self-efficacy between baseline and 6- month follow-up. The Hip School group showed significant improvement in BAS MQ between baseline and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* X-ray-verified hip OA, no walking aid and no joint replacements in the hips or knees.

Exclusion Criteria:

* no OA, joint replacement

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in Hip Osteoarthritis Outcomes Score (HOOS, Swedish version L.K 1.1) | Baseline, 6 month, 12 month
  An instrument for assessing patients' options and limitations associated with their hip problems. The questionnaire consists of 39 items in 5 subscales, pain (P, 9 items), other symptoms including stiffness (S, 5 items), activity limitations daily living (ADL, 17 items), activity limitations recreation and sport (SP, 4 items) and hip-related quality of life (QOL, 4 items).

SECONDARY OUTCOMES:
Change in The Body Awareness Scale Movement Quality (BAS MQ) | Baseline, 6 month
  A physiotherapeutic assessment focusing on body awareness and quality of movements, including quality of everyday functional movements and movement behavior, assessed through observation from a structured movement test.
Change in The Six Minute Walk Test (6MWT). | Baseline, 6 month
  Timed walking tests are used to evaluate functional exercise performance and measure the ability to carry-out the activities of daily life. The total distance in meters covered in 6 minutes was recorded.
Change in Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) | Baseline, 6 month, 12 month
  Assessment of HRQL. SF-36 has two summary scales: a Physical Component Scale, PCS, with four subscales: physical functioning (PF, 10 items), role limitation owing to physical health problems (RP, 4 items), bodily pain (BP, 2 items), general health perception (GH, 5 items) as well as a Mental Component Scale, MCS, with four subscales: vitality (VT, 4 items), social functioning (SF, 2 items), role limitation owing to emotional problems (RE, 3 items) and mental health (MH, 5 items). The scores on all subscales range from 0 to 100, with higher scores indicating better health states.
Change in The Arthritis Self-Efficacy Scale (ASES) | Baseline 6 month, 12 month
  Patient's self-reported judgment of what he/she can do regardless of the degree of functional limitations or skill. The ASES consist of 20 items (3 subscales and a total score) which measures: a person's perceived ability to control pain (SEP, 5 items), self-efficacy to perform functions in daily living (SEF, 9 items) and the self-efficacy to control other symptoms related to chronic disease (SEOS, 6 items). Each item ranges from 10=very uncertain to 100=very certain to accomplish the described task. Each subscale is scored by calculating the mean of the items. A higher score indicates better self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sundén, PhD, Principal Investigator — Lund University

IPD SHARING:
Plan to Share IPD: No
Individual participant data has not been shared with other researchers